CLINICAL TRIAL: NCT06251804
Title: Effectiveness of Short-Foot Exercises in Water and on Land in Pes Planus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-19/03
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water exercise program (Experimental): The treatment program includes in-water exercise program. Participants will be exercised twice a week for six weeks.
  Interventions: Other: Water exercise program
- Land-based-program (Active Comparator): The treatment program includes land-based exercise program. Participants will be exercised twice a week for six weeks.
  Interventions: Other: Land-based-program

INTERVENTIONS:
Other: Water exercise program — The exercise program includes a short foot exercise and will be given in water.
  Arms: Water exercise program
Other: Land-based-program — The exercise program includes a short foot exercise and will be given on land.
  Arms: Land-based-program

SUMMARY:
Pes planus is caused by the elongation of the intrinsic muscles in the medial arch of the foot, causing the arch to approach the ground or the sole of the foot to touch the ground completely.

DETAILED DESCRIPTION:
For this purpose, in this project, the effectiveness of short foot exercises in water and on land will be compared in young adults with pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25
* Having bilateral pes planus
* People with a score of 6 and above on the Foot Posture Index Score
* Individuals with more than 10 millimeters of pronation according to the navicular drop test were included.

Exclusion Criteria:

* Rigid pes planus, hallux valgus, hallux rigidus, epin calcanei
* Lower extremity surgery
* Neurological or orthopedic problems and history of disease
* Regular exercise for the treatment of pes planus in the last three months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index | 6 weeks
  A widely used method to assess foot posture and classify individuals according to different foot types.
  Each criterion is scored on a 5-point scale ranging from -2 to +2.
Navicular Drop Test | 6 weeks
  It is a clinical assessment used to evaluate the degree of foot pronation or flattening of the medial longitudinal arch during weight bearing. It is commonly used to assess foot pronation, especially the vertical displacement of the navicular bone during weight bearing.
Biodex Balance System | 6 weeks
  It is a computerized balance assessment system widely used in clinical and research settings to assess and improve balance and stability. The Biodex Balance System typically consists of a computerized platform with force sensors, visual feedback display and various training modes. It provides quantitative measurements of balance parameters, allowing accurate assessment and monitoring of progress

SECONDARY OUTCOMES:
Pittsburg Sleep Index | 6 weeks
  It is a widely used scale that evaluates sleep quality and disorders related to sleep problems.
  The Pitssburg sleep index includes 19 questions Each question is scored from 0 to 3 points, with a high score indicating poor sleep quality. The scale has a total score with a minimum score of 0 and a maximum score of 21 points

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No